CLINICAL TRIAL: NCT06458218
Title: Population Medicine Multimorbidity Interventions in Xishui on a High-Risk COPD Population with Mental Health Symptoms: a Cluster Randomized Controlled Trial
Brief Title: Impact of Multi-component Interventions on Populations with Mental Health Symptoms and High-risk COPD
Acronym: POPMIX-MH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Collaborators: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Simiao Chen, Professor, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CAMS&PUMC-IEC-2024-043
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-06

CONDITIONS: Multimorbidity; Mental Health Issue; Multi-component Interventions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): We have constructed a pay-for-population mechanism to encourage medical workers caring for population health. We will ask study populations to finish online COPD-SQ questionnaire with notification of his or her COPD high risk status. For high-risk COPD population, we will provide a face-to-face survey and examination, and provide a multi-component intervention at baseline. We give community-based spirometry pulmonary function test and education; If individuals who are COPD patients, they will be encouraged to seek treatment to the superior hospitals. A CBT-based digital health program will be provided. Also health education will be given. Additionally, we provide (1) a digital health intervention programs to smokers; (2) CBT-based health education for the abnormal BMI; (3) active recruitment into National Essential Public Health Program for those with high blood pressure and blood glucose. Intensive follow-ups will be conducted at month 3, 6, 12.
  Interventions: Combination Product: Multi-component Interventions
- Control Arm (No Intervention): Those who are assigned in the control arm, we will ask them to finish the same COPD-SQ online questionnaire with notification of his or her COPD high risk status and a face-to-face survey. No physical examinations, community-based pulmonary function tests will be given.

INTERVENTIONS:
Combination Product: Multi-component Interventions — 1. Community-based spirometry pulmonary function tests and result interpretations and health education for COPD;
  2. A digital health intervention program, EmoEase, for individuals with mental health issues among high-risk COPD population(very familiar with intelligent mobile phone);
  3. NicQuit, digital health intervention to smokers;
  4. Health education to smokers and individuals with mental health issues;
  5. Encouragement to seek professional medication treatment in superior hospitals for spirometry-defined COPD patients;
  6. To actively include individuals whose blood pressure and glucose are higher than the normal value into the National Essential Public Health Service in China;
  7. A CBT-based health education to the BMI abnormal;
  8. Pay-for-performance incentives to medical workers.
  Arms: Intervention arm

SUMMARY:
Study Participants: High-risk COPD population with mental health symptoms, defined as individuals whose score of COPD-SQ ≥ 16, whose age is 35 and above, and whose Warwick-Edinburgh Mental Well-being Scale <45 .

Intervention: We have constructed a pay-for-population mechanism for medical practitioners within the intervention townships to encourage them caring for population health. For study participants in the intervention arm, we will ask them to finish an online COPD-SQ questionnaire with notification of his or her COPD high risk status. For those with high-risk COPD population, we will provide face-to-face survey, simple physical examination, pulmonary function tests, and provide a multi-component intervention at baseline. For high-risk COPD population with mental health issues in the intervention arm, we provide community-based spirometry pulmonary function test (PFT) and education; If individuals whose post-bronchodilator FEV1/FVC<0.7, they will be spirometry-defined COPD patients and will be encouraged to seek treatment and medication to the superior hospitals. A CBT-based digital health intervention program, EmoEase, will be provided to our study participants with an intelligent mobile phone. Also health education in terms of mental health issues will be given. Additionally, we provide (1) a digital health intervention programs to smokers; (2) CBT-based health education for study participants with abnormal BMI; (3) active recruitment into National Essential Public Health Program in China for those with abnormal blood pressure and blood glucose. Intensive follow-ups will be conducted at month 3 (telephone interview), month 6 (face-to-face with full steps of physical examination), and month 12.

Comparison: Those who are assigned in the control arm, we will ask them to finish the same COPD-SQ online questionnaire with notification of his or her COPD high risk status and a face-to-face survey. No physical examinations, community-based pulmonary function tests will be given.

Outcomes: The primary outcomes are PHQ-9 scores for depression symptoms, GAD-7 symptoms for anxiety symptoms, and WEM-WBS score at month 12.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35 and above;
* High-risk COPD population, defined by score of COPD-SQ ≥ 16;
* Mental health issues, defined by WEM-WBS scale < 45;
* Local residents who stay within a township in the previous 3 months and plan to stay within the same township for the next 12 months.

Exclusion Criteria:

* Those who suffer from severe cognitive disorder or total loss of ability of daily living.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7400 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Depression Symptoms | 1 year
  Definition: Emotional disorders, including sadness, loss, and anger; Variable type: Continuous; Measurement: PHQ-9; Introduction to PHQ-9: Patient Health Questionnaire- 9 items (PHQ-9), ranging from 0 to 27, the higher the score, the severer the depression symptoms for the respondents will be.
Anxiety Symptoms | 1 year
  Definition: Unpleasant state of inner turmoil; Variable type: Continuous; Measurement: GAD-7; Introduction to GAD-7: General Anxiety Disorder - 7 (GAD-7), ranging from 0 to 21, the higher the score, the severer the anxiety symptoms for the respondents will be.
Warwick-Edinburgh Mental Well-being Scale, WEM -WBS | 1 year
  Definition: Reflects overall mental health problems; Variable type: Continuous; Measurement: WEMWBS; Introduction to WEMWBS: Warwick-Edinburgh Mental Well-being Scale, ranging from 14 to 70, the lower the score, the worse one's general mental health will be.

SECONDARY OUTCOMES:
Number of chronic diseases controlled | 1 year
  Definition: Among all 7 objectively measured health conditions (depression symptoms, anxiety symptoms, COPD, asthma, BMI, hypertension, type 2 diabetes), number of chronic diseases controlled; Variable type: Counting data; Measurement: Physical examination or validated scales.
Self-rated health status | 1 year
  Definition: General self-assessed health status; Variable type: Continuous; Measurement: EQ-5D scale; Introduction to EQ-5D-5L scale: The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group in 2009 to improve the instrument's sensitivity and to reduce ceiling effects, as compared to the EQ-5D-3L. The scale could be transferred to health utility value, ranging from 0 to 1 continuously. 0 represents death and 1 represents perfect health.
FEV1 measurement | 1 year
  Definition: Forced Expiratory Volume in one second (FEV1); Variable type: Continuous; Measurement: Pulmonary function test, portable spirometry;
mMRC score | 1 year
  Definition: mMRC questionnaire; Variable type: Categorical; Measurement: Respondent's answer to the question; Introduction to mMRC: Modified Medical Research Council, categorical value, level 0 represents a good respiratory condition, while the maximum level 4 represents a very bad respiratory condition.
CAT score | 1 year
  Definition: CAT questionnaire for COPD patients; Variable type: Continuous; Measurement: Respondent's answer to the question; Introduction to CAT questionnaire: COPD Assessment Test (CAT) is a questionnaire for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time. The scope ranges from 0 to 40, the higher the score, the worse the COPD conditions.
COPD Screening | 1 year
  Definition: Have you ever had a pulmonary function test?; Variable type: Binary; Measurement: Respondent's answer to the question;
Self-awareness of COPD | 1 year
  Definition: Have you ever been diagnosed with COPD?; Variable type: Binary; Measurement: Respondent's answer to the question;
COPD-Knowledge | 1 year
  Definition: COPD Knowledge Questionnaire; Variable type: Continuous; Measurement: Respondent's answer to the questions;
Treatment adherence | 1 year
  Definition: Are you currently receiving a COPD treatment plan prescribed by a doctor or other healthcare professional?; Variable type: Binary; Measurement: Respondent's answer to the question;
COPD control | 1 year
  Definition: Has the number of acute exacerbations decreased in the past six months?; Variable type: Binary; Measurement: Respondent's answer to the question;
Blood pressure | 1 year
  Definition: Systolic and diastolic blood pressure (mmHg); Variable type: Continuous; Measurement: Omron portable automatic blood pressure monitor;
Blood Glucose | 1 year
  Definition: Reference standard for average plasma glucose concentration over a period of time; Variable type: Continuous; Measurement: Blood glucose meter;
Waist circumference | 1 year
  Definition: Waist circumference (cm); Variable type: Continuous; Measurement: Soft measuring tape;
BMI | 1 year
  Definition: Body mass index (BMI), weight divided by height squared (kg/m²); Variable type: Continuous; Measurement: Calculation;
Outpatient | 1 year
  Definition: Outpatient visits and type of hospital; Variable type: Count; Measurement: Survey data/insurance/outpatient data;
Inpatient | 1 year
  Definition: Inpatient visits and type of hospital; Variable type: Count; Measurement: Survey data/insurance/outpatient data;
Medical expenditure within a family over the past year | 1 year
  Definition: Healthcare-related expenditures; Variable type: Continuous; Measurement: Survey data/insurance/outpatient/inpatient data;
Productivity Loss | 1 year
  Definition: Productivity loss due to illness or health problems from Working Productivity and Activity Impairment-General Health Chinese version 2.0; Variable type: Continuous; Measurement: Respondent's answer to the question;
  WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes, as follows:
  Questions:
  1. = currently employed
  2. = hours missed due to health problems
  3. = hours missed other reasons
  4. = hours actually worked
  5. = degree health affected productivity while working
  6. = degree health affected regular activities
  Scores:
  Multiply scores by 100 to express in percentages.
  Percent work time missed due to health: Q2/(Q2+Q4)
  Percent impairment while working due to health: Q5/10
  Percent overall work impairment due to health:
  Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4)))x(Q5/10)]
  Percent activity impairment due to health: Q6/10
HBP Screening | 1 year
  Definition: Have you ever had your blood pressure measured by a doctor, nurse, or other healthcare professional?; Variable type: Binary; Measurement: Respondent's answer to the question;
HBP Diagnosis | 1 year
  Definition: Have you ever been diagnosed with hypertension by a doctor?; Variable type: Binary; Measurement: Respondent's answer to the question;
HBP Treatment | 1 year
  Definition: Are you currently taking any antihypertensive medication prescribed by a doctor or other healthcare professional? Variable type: Binary; Measurement: Respondent's answer to the question;
HBP Control | 1 year
  Definition: Blood pressure within the normal range at the end-of-year follow-up; Variable type: Binary; Measurement: Blood pressure measurement
T2DM Screening | 1 year
  Definition: Have you ever had your blood glucose measured by a doctor, nurse, or other healthcare professional?; Variable type: Binary; Measurement: Respondent's answer to the question;
T2DM Diagnosis | 1 year
  Definition: Have you ever been diagnosed with T2DM by a doctor?; Variable type: Binary; Measurement: Respondent's answer to the question;
T2DM Treatment | 1 year
  Definition: Are you currently receiving a type 2 diabetes treatment plan prescribed by a doctor or other healthcare professional?; Variable type: Binary; Measurement: Respondent's answer to the question;
T2DM Control | 1 year
  Definition: Blood glucose within the normal range at the end-of-year follow-up; Variable type: Binary; Measurement: Blood glucose measurement;
Smoking Status | 1 year
  Definition: Do you currently smoke?; Variable type: Binary; Measurement: Respondent's answer to the question;
Smoking Amount | 1 year
  Definition: If yes, how many cigarettes do you smoke per day on average?; Variable type: Count; Measurement: Respondent's answer to the question;
Drinking Status | 1 year
  Definition: Frequency of alcohol consumption in the past 3 months; Variable type: Categorical; Measurement: Respondent's answer to the question;
Sugar Consumption | 1 year
  Definition: Frequency of consumption of sugary foods/drinks; Variable type: Categorical; Measurement: Respondent's answer to the question;
Salted Vegetables Consumption | 1 year
  Definition: Frequency of consumption of salty vegetables; Variable type: Categorical; Measurement: Respondent's answer to the question;
Vegetable Consumption | 1 year
  Definition: Frequency of consumption of vegetable; Variable type: Categorical; Measurement: Respondent's answer to the question;
Physical exercise | 1 year
  Definition: Hours of physical exercise per week; Variable type: Count; Measurement: Respondent's answer to the question;
Smoking Dependence | 1 year
  Fagerström test for nicotine dependence (FTND) is a scale that measures the nicotine dependence of smokers, ranging from 0 to 15, the higher the value, the worse the nicotine dependence will be. Heaviness Index of Smoking (HIS) could also be calculated using part of the scale, ranging from 0 to 6, and higher score means worse nicotine dependence.

CONTACTS AND LOCATIONS:
Overall Officials: Simiao Chen, Ph.D., Principal Investigator — Peking Union Medical College
Locations (1):
- Xishui County, Zunyi, Guizhou, China

IPD SHARING:
Plan to Share IPD: No